CLINICAL TRIAL: NCT03258229
Title: A 8-week, Randomized, Double-blind, Placebo-controlled 2x2 Cross-over Design Human Trial to Evaluate the Efficacy and Safety of Angelica Gigas N. Extract on Improvement of Hyperglycemia
Brief Title: Efficacy and Safety of Angelica Gigas N. Extract on Improvement of Hyperglycemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Wan Chae, Principal Investigator, Clinical Trial Center for Functional Foods, Chonbuk National University Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: WBP-HG-AG2
Record Dates: First submitted 2017-03-09; First posted 2017-08-23 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Hyperglycemia
Keywords: Angelica gigas N. extract; Glucose; Clinical Trial
MeSH Terms: conditions — Hyperglycemia

STUDY DESIGN:
Intervention Model Description: 2×2 cross-over Assignment
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Angelica gigas N. extract (Experimental): capsules(2cap/d, 1,000mg/d) for 8 weeks.
  Interventions: Dietary Supplement: Angelica gigas N. extract
- Placebo (Placebo Comparator): Placebo for 8 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Angelica gigas N. extract — capsules(2cap/d, 1,000mg/d) for 8 weeks.
  Arms: Angelica gigas N. extract
Dietary Supplement: Placebo — Placebo for 8 weeks
  Arms: Placebo

SUMMARY:
This study was conducted to investigate the effects of daily supplementation of Angelica gigas N. extract on improvement of Hyperglycemia .

DETAILED DESCRIPTION:
This study was a 8 weeks, randomized, double-blind, placebo-controlled 2×2 cross-over design human trial. Twenty subjects were randomly divided into Angelica gigas N. extract or a placebo group. Fasting and postprandial glucose profiles during oral glucose tolerance test (OGTT) were assessed before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-80 years with fasting glucose 100-125 mg/dL or 2 hour postprandial glucose 140-199 mg/dl

Exclusion Criteria:

* Weight less than 48 kg or weight decreased by more than 10% within past 3 months
* Hypoglycemic agent, Obesity medicine, Lipid lowering agent within past 6 months or Blood sugar, Obesity and Lipid improvement functional foods within past 2 weeks
* Treated with corticosteroid within past 4 weeks
* Severe cardiovascular disease(Mvocardial infarction, Stroke, etc)
* Renal disease(Heredity hyperlipidemia, Acute/Chronic renal failure, Nephrotic syndrome, etc)
* Rheumatoid arthritis, Autoimmune disease
* Cancer, Respiratory organ disease(Asthma, Chronic obstructive pulmonary disease)
* Allergic or hypersensitive to any of the ingredients in the test products
* History of disease that could interfere with the test products or impede their absorption
* Under antipsychotic drugs therapy within past 2 months
* History of alcohol or substance abuse
* Participation in any other clinical trials within past 2 months
* Laboratory test by show the following results

  * aspartate aminotransferase, alanine aminotransferase > Reference range upper limit treble
  * Serum Creatinine > 2.0 mg/dl
* Pregnancy or breast feeding
* Not Contraception(except: Surgery for female infertility)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-02-09 (Actual); Primary Completion 2017-12-07 (Actual); Study Completion 2017-12-07 (Actual)

PRIMARY OUTCOMES:
Changes of blood glucose during OGTT (oral glucose tolerance test) | 8 weeks
  Changes of fasting and postprandial glucose during OGTT were assessed before and after the intervention.

SECONDARY OUTCOMES:
Changes of blood insulin during OGTT | 8 weeks
  Changes of blood insulin during OGTT were assessed before and after the intervention.
Changes of Homeostatic model assessment-insulin resistance | 8 weeks
  Changes of physiological parameter{Homeostatic model assessment-insulin resistance(mg/dl)} were assessed before and after the intervention
Changes of Homeostatic model assessment-beta-cell | 8 weeks
  Changes of physiological parameter{Homeostatic model assessment-beta-cell(mg/dl)} were assessed before and after the intervention
Changes of HbA1c | 8 weeks
  Changes of HbA1c(%) were assessed before and after the intervention
Changes of Adiponectin, Leptin | 8 weeks
  Changes of Adiponectin and Leptin(ng/ml) were assessed before and after the intervention
Changes of lipid profile | 8 weeks
  Changes of lipid profile were assessed before and after the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Center for Functional Foods; Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided